CLINICAL TRIAL: NCT06168877
Title: Use of Integrated PET/CT as a First Line Staging and Re-staging Technique in Oncologic Patient.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PET/TC and TCMDC
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Execution of 18F-FDG PET/CT and contrast-enhanced CT scan. — PET/CT, contrast-enhanced CT and contrast-enhanced PET/CT+CT performed in a single examination session (single staging) in cancer patients (patients suffering from lymphoma and lung cancer).

SUMMARY:
Positron emission tomoscintigraphy (PET) and contrast computed tomography (CTmdc) are diagnostic methods widely used in the staging and restaging of neoplastic diseases. In recent years, PET tomographs have been implemented, integrating a CT scanner into the PET tomograph (PET/CT): these tomographs are able to simultaneously acquire the function/metabolism study (PET) and the morgfostructural study (CT).

Numerous clinical studies have demonstrated the added diagnostic value of PET/CT compared to PET with consequent effect on the choice of treatment type. In addition to the potential clinical value deriving from the simultaneous execution of the two diagnostic methods, it is necessary to consider the possibility of a reduction in indirect costs deriving from the reduction of days of work lost and costs related to transport, both for the patient and for any companions.

The aims of this multicenter observational study are:

1. evaluate the diagnostic accuracy of PET/CT, contrast-enhanced CT and contrast-enhanced PET/CT+CT performed in a single examination session (single staging) in cancer patients (patients suffering from lymphoma and lung cancer).
2. evaluate any psychological, quality of life and economic benefits deriving from carrying out the two diagnostic procedures in a single examination session.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from lung cancer or lymphoma in which the two diagnostic investigations mentioned (PET and contrast-enhanced CT) are part of the routine diagnostic-therapeutic program of the disease in question;
* Patients suffering from lung cancer will be in the stage of primary neoplasm staging;
* Patients suffering from lymphoma will be evaluated both in the disease staging phase at onset and re-evaluation after radio-chemotherapy treatment.

Exclusion Criteria:

* Patients with contraindications to performing investigations with contrast medium.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients suffering from lymphoma or lung cancer undergoing PET/CT and contrast-enhanced CT in a single examination session.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-10-21 (Actual); Primary Completion 2014-07-03 (Actual); Study Completion 2014-07-03 (Actual)

PRIMARY OUTCOMES:
Use of PET/CT, contrast-enhanced CT and contrast-enhanced PET/CT+CT performed in a single examination session in cancer patients. | 5 years
  Use of PET/CT, contrast-enhanced CT and contrast-enhanced PET/CT+CT performed in a single examination session in cancer patients in terms of diagnostic accuracy, quality of life and economic aspects.

IPD SHARING:
Plan to Share IPD: No